CLINICAL TRIAL: NCT01502670
Title: A Pilot Study of the Utility of the Novel Amino Acid Radiotracer Anti-[18 F]FACBC for the Noninvasive Imaging of Lung Nodules
Brief Title: Amino Acid Tracer (FACBC) Positron Emission Tomography for Lung Nodule
Acronym: SPN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Nihon Medi-Physics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, David M. Schuster, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00006621; 14701 (Other: Other)
Record Dates: First submitted 2011-12-21; First posted 2012-01-02 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Lung Cancer
Keywords: Pulmonary nodules
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lung Nodule (Experimental)
  Interventions: Drug: 18F-FACBC Radiotracer

INTERVENTIONS:
Drug: 18F-FACBC Radiotracer — Test radiotracer uptake in lung nodule
  Other Names: Radiotracer

SUMMARY:
This study will look at how the [18]FACBC goes into the lung nodules. This will hopefully lead to the development of better imaging techniques to look at lung nodules. [18]FACBC is not approved by the FDA (Food and Drug Administration). This study will help to determine if it should be approved by the FDA.

DETAILED DESCRIPTION:
This is a study that will test a compound (chemical substance) that has a small amount of radioactivity attached to it. This substance has a natural tendency to go to tumor cells, as has been shown in the detection and staging of prostate cancer and for brain tumors. In this study we are going to test this new substance in patients with lung nodules. Lung nodules are a common finding. It is very important to non-invasively determine whether the nodule is cancer or not, as early cancer detection and treatment may cure the disease. The substance is called [18]FACBC and it is given in the form of an injection into a vein. After the substance reaches the lung nodules, scans called PET or Positron Emission Tomography, are done. This is similar to having CAT scans or x-rays. Usually a compound called [18]FDG is used for PET scans but this substance often goes to inflammatory tissues as well. This new substance does not significantly go to inflammatory tissues, and may allow tumors in the lungs to be better identified.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients with a history of cancer who have a solitary pulmonary nodule between 1-3 cm in short axis with clinical and CT characteristics warranting surgical removal (see below).
3. Clinical, laboratory, or diagnostic imaging findings on CT or 18F-FDG PET-CT do not suggest the possibility of the SPN being part of a metastatic process.
4. Ability to lie still for PET scanning
5. Patients must be able to provide written informed consent.

Exclusion Criteria:

1. Age less than 18.
2. Active carcinoma with known metastatic disease.
3. Size of primary lesion less than 1 cm or greater than 3 cm
4. Not a candidate for surgical resection or biopsy based upon clinical condition or discovery of metastatic disease which would preclude surgical therapy.
5. Inability to lie still for PET scanning
6. Cannot provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Correlation of Radiotracer Uptake with Histology | Typically 1-2 months
  We will correlate radiotracer uptake with histology results

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Amzat R, Taleghani P, Miller DL, Beitler JJ, Bellamy LM, Nye JA, Yu W, Savir-Baruch B, Osunkoya AO, Chen Z, Auffermann WF, Goodman MM, Schuster DM. Pilot study of the utility of the synthetic PET amino-acid radiotracer anti-1-amino-3-[(18)F]fluorocyclobutane-1-carboxylic acid for the noninvasive imaging of pulmonary lesions. Mol Imaging Biol. 2013 Oct;15(5):633-43. doi: 10.1007/s11307-012-0606-7. PMID 23595643